CLINICAL TRIAL: NCT04359485
Title: Use Of A Novel Quantitative Tool For Evaluation of Pseudo- Acanthosis Nigricans: Acanthosis Nigricans Area And Severity Index
Brief Title: New Score for Pseudo- Acanthosis Nigricans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Principal Investigator, Kasr El Aini Hospital
Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EgyANASI
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pseudo Acanthosis Nigricans
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glycolic acid peel (Experimental)
  Interventions: Procedure: Glycolic acids peel 70%
- Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Procedure: Glycolic acids peel 70% — Glycolic acid peel 70% applied in 3 coats medium depth
  Arms: glycolic acid peel
Other: Saline — Sodium chloride
  Arms: Saline

SUMMARY:
Each side of the neck pseudo acanthosis nigricans was randomized in to either receiving glycolic acid peel or saline. Evaluation was done at baseline and after 3 sessions 2 weeks apart by percentage involvement and by ANASI score

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate severity
* age > 18 years old

Exclusion Criteria:

* Pregnant and lactating patients,
* patients with systemic diseases as connective tissue disease, diabetes,
* skin infection
* use of immunosuppressive drugs
* Susceptibility for post peel hazards as hyperpigmentation
* scarring and keloidal tendency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Percentage involvement | 6 months to 1 year
  Degree of severity expressed as a percentage
Acanthosis Nigricans Area and Severity Index score | 6 months to 1 year
  New Score calculating severity and area as a number minimum value is 0 and maximum value is 40 the higher the number of the score the worse the affection

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy university hospital, Faulty of medicine,Cairo university, Cairo, Egypt